CLINICAL TRIAL: NCT03124394
Title: Prospective Intraperitoneal Chemotherapy in Carcinomatosis Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Other Study IDs: Carcinomatosis studyWinterthur
Record Dates: First submitted 2017-04-06; First posted 2017-04-21 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRS and intraoperative chemotherapy: Patients receiving cytoreductive surgery and intraoperative chemotherapy (HIPEC/PIPAC)

SUMMARY:
Evaluation of clinical outcome and economical aspects in the treatment of patients with peritoneal carcinomatosis.

DETAILED DESCRIPTION:
Peritoneal carcinomatosis is a dooming finding with no hope for cure and a steadily decrease in quality of life. Cytoreductive surgery with intraperitoneal chemotherapy (CRS HIPEC) offers a small but proven chance for cure. The implementation of a CRS HIPEC and PIPAC programme in a Swiss tertiary care hospital is evaluated.

When a patient is deemed non resectable, pressurized intraperitoneal aerosol chemotherapy (PIPAC) administered laparoscopically may confer effective palliation.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women >18 years
* Tumour board decision for CRS and intraoperative chemotherapy

Exclusion Criteria:

* Missing Tumour board decision for CRS and intraoperative chemotherapy
* Pregnancy
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peritoneal carcinomatosis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative surgical complications | 90 days
  Reporting and grading of postoperative surgical complications (according to Dindo)
Rehospitalisation | 90 days
  Rehospitalisation: (yes/no), time frame, cause of rehospitalisation
Disease-free survival | 5 years
  Time to recurrence measured since diagnosis/Intervention (in months)
Overall Survival | 5 years
  All cause mortality since diagnosis/Intervention (in months)

SECONDARY OUTCOMES:
Measurement of quality of life | 5 years
  Validated measurements of health-related quality of life according to the EORTC manual in terms of general quality of life: EORTC-QLQ30; disease-specific quality of life: EORTC-CR29 (colorectal cancers), and health-utility (EQ-5D).
Cost | 90 days
  At the level of individual patient Cost in terms of hospital charges and expenses in Swiss Francs
Revenues | 90 days
  At the level of individual patient Revenues in Swiss Francs as billed according to the DRG and case-mix index
Cost-utility analysis | 90 days
  Calculation and comparison of QUALY (quality-adjusted life years derived from EQ-5D) for competing treatment strategies taking advantage of published figures and own data, e.g. cost of a systemic palliative chemotherapy compared to cost of an intraperitoneal chemotherapy
Cost-effectiveness | 90 days
  Aggregation of costs, charges, and revenues for the whole series and comparison with alternative treatment option as clinically relevant, chemotherapy alone and palliative surgery alone.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Adamina, Prof/MD/MSc, Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided